CLINICAL TRIAL: NCT03426514
Title: Single-center Prospective Randomized Controlled Study of the Three-port Laparoscopic Surgery Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Brief Title: Three-port Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, Chief Physicion, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-TLSC-2018
Record Dates: First submitted 2018-01-31; First posted 2018-02-08 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Laparoscopic surgery; Three-port
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-port Laparoscopic Surgery (Experimental): Patients with colorectal cancer undergo three-port laparoscopic surgery.
  Interventions: Procedure: Three-port Laparoscopic Surgery
- Conventional Laparoscopic Surgery (Experimental): Patients with colorectal cancer undergo conventional laparoscopic surgery（4 or more ports）.
  Interventions: Procedure: Conventional Laparoscopic Surgery

INTERVENTIONS:
Procedure: Three-port Laparoscopic Surgery — Patients undergo three-port laparoscopic surgery. The surgery will be completed by a surgeon and a camera-person without another assistant. The surgeon will adjust surgical position to expose the operative field with the help of gravity. All the orther operative procedures are the same as conventional laparoscopic surgery.
  Arms: Three-port Laparoscopic Surgery
Procedure: Conventional Laparoscopic Surgery — Patients undergo conventional laparoscopic surgery（4 or more ports）.The surgery will be routinely completed by a surgeon，a camera-person and another assistant to provide counter-traction.
  Arms: Conventional Laparoscopic Surgery

SUMMARY:
This study is designed to evaluate the short-term and long-term results after three-port laparoscopic surgery for colorectal cancer（TLSC） compared with conventional laparoscopic surgery for colorectal cancer（CLSC）.

DETAILED DESCRIPTION:
At present，surgical treatments is the main means to cure colorectal cancer（CRC）.The use of four or more ports has been routine in most laparoscopic colorectal resections. However，the drawbacks are the need for added manpower, consisting of another assistant to provide counter-traction, as well as costs and the unaesthetic effects of additional ports. In order to minimize surgical trauma, improve cosmesis ,reduce manpower，single-incision laparoscopic surgery (SILS) is attracting increasing attention. But it is challenging and highly demanding techniques. Becoming proficient at three-port laparoscopic surgery can make the transition to SILS more nature.Few studies about three-port laparoscopic surgery for colorectal cancer（TLSC） have been reported currently.More studies, especially large-scale, randomized controlled trials are needed to establish the best indications for TLSC. This is a single-center, open-label, non-inferiority, randomized controlled trial. A total of 282 eligible patients will be randomly assigned to TLSC group and CLSC group at a 1:1 ratio. It will provide valuable clinical evidence for the objective assessment of the the feasibility, safety, and potential benefits of TLSC compared with CLSC.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) <30 kg/m2
* Tumor located in colon and high rectum (the lower border of the tumor is above the peritoneal reflection)
* Pathological colorectal carcinoma
* Clinically diagnosed cT1-4aN0-2 M0 lesions according to the 7th Edition of AJCC Cancer Staging Manual with or without neoadjuvant therapeutic history
* ECOG score is 0-1
* ASA score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Previous gastrointestinal surgery
* History of inflammatory bowel disease
* History of familial adenomatous polyposis（FAP）
* Pregnant woman or lactating woman
* Severe mental disease
* Intolerance of surgery for severe comorbidities
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by colorectal cancer
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Early morbidity rate | 30 days after surgery
  morbidity rate 30 days after surgery

SECONDARY OUTCOMES:
Operative time | intraoperative
  Operative time（minutes）
Intraoperative blood loss | intraoperative
  Estimated blood loss（milliliters，ml）
Lymph node detection | 14 days after surgery
  Lymph nodes harvested（numbers）
Proximal resection margin | 14 days after surgery
  Length of proximal margin （centimeters，cm）
Distal resection margin | 14 days after surgery
  Length of distal margin （centimeters，cm）
Length of stay | 1-14 days after surgery
  Duration of hospital stay（days after surgery）
Postoperative recovery course | 1-14 days after surgery
  Time to first ambulation, flatus, liquid diet and soft diet （hours after surgery）
Pain score | 1-3 days after surgery
  Postoperative pain is recorded using the visual analog scale (VAS) pain score （0-10 points）tool on postoperative day 1, 2, 3 and the day of discharge
3-year disease free survival rate | 36 months after surgery
  3-year disease free survival rate
5-year overall survival rate | 60 months after surgery
  5-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tawfik Amin A, Elsaba TM, Amira G. Three ports laparoscopic resection for colorectal cancer: a step on refining of reduced port surgery. ISRN Surg. 2014 Mar 12;2014:781549. doi: 10.1155/2014/781549. eCollection 2014. PMID 25006515
- [Background] Seow-En I, Tan KY, Mohd Daud MA, Seow-Choen F. Traditional laparoscopic colorectal resections can be performed effectively using a three-port technique. Tech Coloproctol. 2011 Mar;15(1):91-3. doi: 10.1007/s10151-010-0660-6. Epub 2011 Jan 14. No abstract available. PMID 21234638